CLINICAL TRIAL: NCT02581813
Title: Effects of a Weight Management Intervention With Increased Dairy Intake on Body Composition and Bone Health in Overweight and Obese Girls.
Brief Title: Does Dairy Benefit Bone & Body Composition in Overweight Girls Undergoing a Weight Management Program?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Andrea Josse, Assistant Professor, Department of Kinesiology, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 14-284
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Overweight; Obesity; Children
Keywords: Bone health; Body composition; Dairy foods; Exercise; inflammation; nutrition intervention; weight management
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- RDa (Recommended dairy group) (Experimental): 4 servings of dairy per day + exercise (3 times per week with combination of aerobic and resistance exercise).
  Interventions: Behavioral: I.D.E.A.L. for Adolescents Study - Higher Dairy
- LDa (Low dairy group) (Experimental): 0-1 serving of dairy per day + exercise (the same as the RDa group)
  Interventions: Behavioral: I.D.E.A.L. for Adolescents Study - Lower Dairy
- GCon (growth controls) (No Intervention): This no-intervention group will serve as the control to account for growth during the study.

INTERVENTIONS:
Behavioral: I.D.E.A.L. for Adolescents Study - Higher Dairy — 12 weeks diet and exercise intervention characterized by higher dairy consumption (4 servings per day) and exercise 3 times per week
  Arms: RDa (Recommended dairy group)
Behavioral: I.D.E.A.L. for Adolescents Study - Lower Dairy — 12 weeks diet and exercise intervention characterized by lower dairy consumption (0-1 serving per day) and exercise 3 times per week
  Arms: LDa (Low dairy group)

SUMMARY:
The purpose of this study is to examine whether increased dairy intake, at the level recommended by Canada's Food Guide, combined with healthy eating and exercise, will improve body composition and bone turnover over 12 weeks in overweight and obese girls.

DETAILED DESCRIPTION:
Three groups will participate in this study. Participants must be low dairy consumers (0-1 svgs/d) and do little to no structured physical activity at study entry. Each participant will be assigned to a group; one of two experimental groups or a control group. The two intervention groups will differ only in the amount of dairy consumed (4 svgs vs. 0-1 svg/d). Both will undergo the same exercise program (3x/wk) and will be counseled on healthy eating by a trained nutritionist-dietitian every month. The control group will be tested at the beginning and end of the study to help account for any growth-related changes during the study but will not receive any formal intervention. In each group, the investigators will assess body composition (muscle mass, fat mass, % body fat and regional fat mass) and bone (bone turnover markers). The investigators will also measure various metabolic and inflammatory markers, hormones as well as dietary intake, strength and fitness.

This study will determine whether increased intake of dairy products improve bone and body composition during a 12-week weight management intervention. The investigators expect the two groups participating in the intervention to show significant changes in body weight and body composition and greater gains in fitness compared to the control group. The investigators expect those consuming dairy to show greater improvements in body composition and bone health compared to those not consuming added dairy. The investigators also anticipate better vitamin D status and less whole-body inflammation in those consuming dairy. Both intervention groups should show improvements in fasting insulin, glucose and cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* at or above the age appropriate cut-offs for overweight (OW) or obese (OB) on WHO growth charts: ≥85-97% for OW and >97% for OB for BMI
* between 10 and 18 years old
* menarcheal
* low dairy consumers (0-2 svgs/d and <700 mg Ca/d measured by baseline FFQ)
* otherwise healthy (i.e. no diagnosed disease or illness)
* lower levels of physical activity (0-2 times/week)
* no allergy to dairy foods or diagnosed lactose intolerance
* not on medications related to a chronic condition or that affect bone health

Participants will be excluded from participation in the study if they do not meet one or more of the above inclusion criteria.

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2016-05; Primary Completion 2018-10 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in lean mass | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  body composition: lean mass (kg)
Change in fat mass | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  body composition: fat mass (kg)
Change in % body fat | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  body composition: % body fat

SECONDARY OUTCOMES:
Change in TNF-α | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  inflammatory marker: tumor necrosis factor alpha (TNF-α; ng/L)
Change in IL-6 and IL-1β | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  inflammatory markers: Interleukin 6 (IL-6; ng/L), interleukin 1 beta (IL-1β; ng/L)
Change in Leptin | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  adipokine: leptin (mg/L)
Change in Adiponectin | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  adipokine: adiponectin (mg/L)
Change in lipids | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  cardiometabolic risk: lipids (triglycerides, LDL, HDL, total cholesterol; mmol/L)
Change in glucose | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  cardiometabolic risk: glucose (mmol/L)
Change in insulin | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  cardiometabolic risk: insulin (pmol/L)
Change in 25OHD | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  hormone: 25-hydroxyvitamin D (25OHD nmol/L)
Change in PTH | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  hormone: parathyroid hormone (PTH pmol/L)
Changes in fitness | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  cardiovascular fitness and response to exercise (heart rate (HR; bpm) , oxygen consumption (VO2 max) using a progressive exercise test to exhaustion.
Change in P1NP | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  bone turnover biomarker: P1NP (ug/L)
Change in CTx | 3 times during the study (week 0 pre-intervention; week 12 post-intervention; week 24 follow-up)
  bone turnover biomarker: CTx (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Josse, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No